CLINICAL TRIAL: NCT05271630
Title: Multiple Myeloma Outcomes Based on Maintenance Therapy Post Autologous Stem Cell Transplant
Status: Active, not recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Adaptive Biotechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: MCC-20816
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Adjuvants, Immunologic; Proteasome Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Minimal Residual Disease (MRD) testing by Clonoseq will be performed in the peripheral blood of the patients at the same time points that MRD testing will be done in the bone marrow in addition to at 6 and 18 months.
  Investigators will examine the impact gut microbiota on MRD status and racial ethnic differences in study population. Stool samples will be collected at baseline and 1- and 2-years post Autologous Stem Cell Transplant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single Maintenance After Autologous Stem Cell Transplant: Prospectively enrolled cohort of patients receiving single maintenance therapy with an immunomodulatory drug after Autologous Stem Cell Transplant for Multiple Myeloma
  Interventions: Other: Autologous Stem Cell Transplant; Drug: Immunomodulatory Agent
- Double Maintenance After Autologous Stem Cell Transplant: Prospectively enrolled cohort of patients receiving double maintenance therapy with the combination of an immunomodulatory drug and a proteasome inhibitor after Autologous Stem Cell Transplant for Multiple Myeloma.
  Interventions: Other: Autologous Stem Cell Transplant; Drug: Immunomodulatory Agent; Drug: Proteasome Inhibitor

INTERVENTIONS:
Other: Autologous Stem Cell Transplant — This observational study will compare outcomes of prospectively enrolled ASCT recipients receiving Single agent vs doublet maintenance chemotherapy post ASCT
Drug: Immunomodulatory Agent — ASCT recipients receiving maintenance therapy consisting of an Immunomodulatory agent (IMID) after ASCT transplant
Drug: Proteasome Inhibitor — ASCT recipients receiving maintenance therapy with a proteasome inhibitor in combination with an immunomodulatory drug after ASCT transplant
  Groups: Double Maintenance After Autologous Stem Cell Transplant

SUMMARY:
The purpose of the study is to determine outcomes for Multiple Myeloma patients on maintenance single agent vs. doublet (IMiD + PI) combination chemotherapy post Autologous Stem Cell Transplant (ASCT).

DETAILED DESCRIPTION:
This non-interventional, cohort prospective research study will assess outcomes for Multiple Myeloma patients on maintenance single agent vs. doublet (IMiD + PI) combination chemotherapy post ASCT.

ELIGIBILITY:
Inclusion Criteria:

* All MM patients (18 years or greater) receiving autologous transplantation given as first line therapy (Melphalan at least 140 mg/m2) will be screened and enrolled in the study if they qualify and willing to participate.
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
* Histologically confirmed diagnosis of multiple myeloma.
* Received high dose melphalan (≥ 140 mg/m2) followed by ASCT based on the institutional guidelines and within +60 and +180 after ASCT at the time of maintenance initiation.
* Disease status must be very good partial response (VGPR), complete remission (CR), or stringent complete remission (sCR) per IMWG response criteria at time of study entry.
* Measurable disease at diagnosis per IMWG criteria serum M spike ≥ 1g/dL, or Urine M protein ≥ 200 mg/24h or involved free light chain ≥ 100 mg/L with an abnormal ratio.
* Patients must have the Clonoseq ID sample showing a trackable clone in bone marrow.

Exclusion Criteria:

* Patients who have purely non-secretory multiple myeloma (i.e., the absence of a measurable protein in serum by electrophoresis and immunofixation and the absence of Bence-Jones protein in the urine defined by use of electrophoresis and immunofixation)
* Prior evidence of disease progression
* Patients who have other malignancy associated with a high risk of progression in the next 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Myeloma patients receiving treatment at Moffitt Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
MRD conversion rate | At 1 year after transplant
  To determine rate of MRD conversion (positive to negative) in MM patients receiving an immunomodulatory drug in combination with a proteasome inhibitor as maintenance therapy 1-year post transplant.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) at 1 Year | At 1 Years
  PFS is defined as time from transplant to disease progression, death or last follow-up date, whichever comes first. PFS will be estimated by Kaplan-Meier method and 95% confidence interval
Progression Free Survival (PFS) at 2 Years | At 2 years
  PFS is defined as time from transplant to disease progression, death or last follow-up date, whichever comes first. PFS will be estimated by Kaplan-Meier method and 95% confidence interval
MRD by NGS Clonoseq testing | At 2 years
  MRD testing by NGS Clonoseq in peripheral blood of participants and correlate with same testing in bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Doris Hansen, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Clinical Trial Search — https://moffitt.org/clinical-trials-research/clinical-trials/